CLINICAL TRIAL: NCT00848016
Title: A Phase II Study of the Orally Administered Negative Enantiomer of Gossypol (AT-101) in Patients With Advanced Adrenocortical Carcinoma (ACC)
Brief Title: Gossypol Acetic Acid in Treating Patients With Recurrent, Metastatic, or Primary Adrenocortical Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01160; MC0771; 8035; CDR0000635024; N01CM00070 (NIH); N01CM00038 (NIH)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Adrenocortical Carcinoma; Stage III Adrenocortical Carcinoma; Stage IV Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — gossypol acetic acid

ARMS (1):
- Treatment (R-(-)-gossypol acetic acid) (Experimental): Patients receive 20mg oral R-(-)-gossypol acetic acid once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: R-(-)-gossypol acetic acid

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid — Participants take 20mg oral R-(-)-gossypol acetic acid once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: AT-101

SUMMARY:
This phase II trial is studying how well gossypol acetic acid works in treating patients with recurrent, metastatic, or primary adrenocortical cancer that cannot be removed by surgery. Drugs used in chemotherapy such as gossypol acetic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of patients with recurrent, metastatic, or primary unresectable adrenocortical carcinoma who achieve an objective response to R-(-)-gossypol acetic acid.

SECONDARY OBJECTIVES::

I. To evaluate the safety of this drug in these patients. II. To determine the progression-free and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive oral R-(-)-gossypol acetic acid once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adrenocortical carcinoma

  * Recurrent, metastatic, or primary unresectable disease
* Measurable disease, defined as ≥ 1 lesion accurately measured in ≥ 1 dimension as ≥ 2.0 cm by conventional techniques or ≥ 1.0 cm by spiral CT scan
* No adrenocortical tumors that, in the Principal Investigator's opinion, are potentially resectable by surgical excision alone
* No symptomatic or progressive brain metastases

  * Patients with treated brain metastases ≥ 6 months prior to study who are clinically and radiographically stable or improved and are off steroids are eligible
  * Must undergo an MRI of the brain or CT scan of the head with contrast ≤ 4 weeks prior to study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy ≥ 12 weeks
* White blood cell count (WBC) ≥ 3,000/mm3
* Absolute neutrophil count (ANC) ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 1.7 mg/dL or creatinine clearance ≥ 40 mL/min
* Able to take oral medications on a regular basis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for ≥ 1 month after completion of study treatment
* No HIV positivity
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No condition or disease that significantly affects gastrointestinal (GI) function or impairs the ability to swallow and retain oral medications including, but not limited to, any of the following:

  * GI tract disease or a requirement for IV alimentation
  * Prior resection of the stomach or small bowel or surgical procedures affecting absorption
  * Active peptic ulcer disease
  * Malabsorption syndrome
  * Ulcerative colitis
  * Inflammatory bowel disease
  * Partial or complete small bowel obstruction
* No other malignancy within the past 2 years except nonmelanoma skin cancer or in situ cervical cancer
* No symptomatic hypercalcemia > grade 2
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to R-(-)-gossypol acetic acid
* Fully recovered from prior surgical procedures and recovered to ≤ grade 1 from adverse events due to previous treatments
* No prior racemic gossypol or R-(-)-gossypol acetic acid
* More than 4 weeks since prior chemotherapy, biologic therapy, major surgery, or radiotherapy (≥ 6 weeks for carmustine or mitomycin C)
* Prior and concurrent mitotane and ketoconazole allowed for patients with hormonal excess
* More than 4 weeks since prior and no concurrent treatment with another investigational agent
* No concurrent prophylactic use of hematopoietic growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], interleukin-11) during the first course of study treatment
* Not requiring routine use of platelet transfusions to maintain ANC or platelet count above required thresholds

Exclusion Criteria:

* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Menefee, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened on 3/17/2009 and accrued 29 participants before being permanently closed 8/03/2011.
Pre-assignment Details: All 29 participants are off treatment, and all participants are evaluable for response and for adverse responses.
Period: Overall Study
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 50 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Achieve a Confirmed Objective Response to Treatment, Either Partial Response (PR) or Complete Response (CR) as Defined by Response Evaluation Criteria In Solid Tumors (RECIST) Criteria
Description: In order for a patient to be a confirmed objective responder, they must achieve a PR or CR on consecutive evaluations, at least 4 weeks apart. The proportion of patients who achieve a confirmed objective response to treatment will be estimated by the standard binomial estimator, i.e., the number of successes divided by the total number of evaluable patients.
  Complete Response (CR): Disappearance of all target lesions and normalization of tumor biomarkers.
  Partial Response (PR): At least a 30% decrease in the sum of the longest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 29
percentage of participants | 0 [NA to NA] — No confidence interval was estimated due to a lack of response.

2. Secondary Outcome: Overall Survival
Description: The overall survival time is defined as the time from registration to date of last follow-up or death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to date of last follow-up or death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 29
months | 8.5 [5.0 to 9.8]

3. Secondary Outcome: Progression-free Survival
Description: The progression-free survival is defined as the time from registration to the date of progression or death, whichever comes first. The distributions of progression-free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to progression or death, whichever occurs first, up to 2 years.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 29
months | 1.9 [1.8 to 2.0]

ADVERSE EVENTS:
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Serious Adverse Events (participants affected / at risk) | 11/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol Acetic Acid) (N=29)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Cardiac troponin T increased (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol Acetic Acid) (N=29)
Hemoglobin decreased (Blood and lymphatic system disorders) | 21 (57)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (20)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 9 (18)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (12)
Vomiting (Gastrointestinal disorders) | 4 (6)
Chills (General disorders) | 1 (2)
Edema limbs (General disorders) | 2 (5)
Fatigue (General disorders) | 8 (13)
Fever (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 7 (12)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Bilirubin increased (Investigations) | 2 (2)
Cardiac troponin I increased (Investigations) | 1 (1)
Cardiac troponin T increased (Investigations) | 3 (4)
Creatinine increased (Investigations) | 5 (7)
Laboratory test abnormal (Investigations) | 3 (3)
Leukocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 9 (17)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Taste alteration (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3)
Flushing (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less